CLINICAL TRIAL: NCT01797887
Title: Diet and Lifestyle Modification in Mothers With Burnout-Syndrome: Ayurvedic Versus Conventional Standard Counseling - A Randomized Controlled Clinical Pilot Study
Brief Title: Ayurvedic Versus Conventional Counseling in Mothers With Burnout-Syndrome
Acronym: VEDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other); European Association for Ayurveda Therapists, Germany (VEAT) (Unknown)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med. Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VEDA-Trial
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Burnout-Syndrome
Keywords: Burnout-Syndrome; Ayurveda; Ayurvedic; Traditional Indian Medicine; CAM; Whole Medical System; Diet and Lifestyle Counseling
MeSH Terms: conditions — Burnout, Psychological | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ayurveda (Experimental): Ayurveda Diet and Lifestyle Counseling
  Interventions: Behavioral: Diet and Lifestyle Counseling
- Conventional (Active Comparator): Standard Conventional Diet and Lifestyle Counseling
  Interventions: Behavioral: Diet and Lifestyle Counseling

INTERVENTIONS:
Behavioral: Diet and Lifestyle Counseling — Diet and Lifestyle Counseling

SUMMARY:
Aim of this study is to evaluate the effectiveness of Ayurvedic diet and lifestyle counseling compared to conventional standard diet and lifestyle counseling in outpatient mothers with burnout-syndrome.

DETAILED DESCRIPTION:
Ayurveda is a traditional Indian medicine: as a whole medical system it consists of diagnostic procedures and complex treatments. Ayurveda-treatment is based on Ayurvedic diagnosis and has a special focus on lifestyle and nutritional counseling, based on the individual constitution of the patient. Ayurvedic counseling can easily be followed by the patients in their day-to-day life and is an inexpensive way of self-care. In Ayurveda it is often used for the treatment of burnout-syndrome. However, no systematic data is available on its effectiveness in comparison to conventional standard diet and lifestyle counseling. The aim of this study is to evaluate the effectiveness of Ayurvedic diet and lifestyle counseling compared to conventional standard diet and lifestyle counseling in outpatient mothers with burnout-syndrome.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age between 18 and 50
* mother of ≥ 1 child ≤ 12 years of age
* job, education or studies ≥ 20 hours per week
* subjective feeling of physical and mental exhaustion since ≥ 3 month
* ≥ 18 points in the MBI Subscale "emotional exhaustion" at screening

Exclusion Criteria:

* change of psychotropic drug medication ≤ 6 weeks before inclusion
* pregnancy or breastfeeding
* pre-diagnosed major depression
* serious chronic co-morbidity (e.g. CHF NYHA IV)
* serious acute somatic health conditions
* intake of opiods
* simultaneous participation in other trials
* praticipation in other trials during ≤ 6 month before inclusion

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maslach-Burnout-Inventory (MBI) | 3 month

SECONDARY OUTCOMES:
Maslach-Burnout-Inventory (MBI) | 6 month
Cohen Perceived Stress Scale (CPSS) | 3 and 6 month
Hospital Anxiety and Depression Scale (HADS-D) | 3 and 6 month
SF-36 | 3 and 6 month
Aspects of Spirituality (ASP) | 3 and 6 month
Pittsburgh Sleep Quality Index (PSQI) | 3 and 6 month

OTHER OUTCOMES:
Qualitative Interviews | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, MD, Principal Investigator — Charité Medical University Berlin, Germany
Locations (1):
- Immanuel Hospital Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Kessler CS, Eisenmann C, Oberzaucher F, Forster M, Steckhan N, Meier L, Stapelfeldt E, Michalsen A, Jeitler M. Ayurvedic versus conventional dietary and lifestyle counseling for mothers with burnout-syndrome: A randomized controlled pilot study including a qualitative evaluation. Complement Ther Med. 2017 Oct;34:57-65. doi: 10.1016/j.ctim.2017.07.005. Epub 2017 Jul 16. PMID 28917376
- See also: Immanuel Hospital Berlin, Germany — http://www.naturheilkunde.immanuel.de
- See also: Cahrité Medical University Berlin, Germany — http://www.charite.de